CLINICAL TRIAL: NCT06897059
Title: Effectiveness of Smartphone Application (Vuka+) for Adherence Support in Adolescent Girls and Young Women -Type I Hybrid Implementation Trial
Brief Title: Effectiveness of Smartphone Application for Adherence Support (Vuka+)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: CONRAD (Other); Desmond Tutu Health Foundation (Other); Florida State University (Other); University of North Carolina, Chapel Hill (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); Gilead Sciences (Industry); Old Dominion University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D21-152
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-01

CONDITIONS: Adherence, Medication; Smartphone Application
Keywords: PrEP; HIV; smartphone
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): Participants received PrEP standard of care counselling per country guidelines
- Vuka+ App (Experimental): Participants downloaded and accessed the Vuka+ application in addition to receiving PrEP standard of care counseling.
  Interventions: Other: Vuka+ application

INTERVENTIONS:
Other: Vuka+ application — The Vuka+ smartphone app included PrEP daily reminders, tracking for pill taking, resources for sexual reproductive health including quizzes and articles, and chat access to other Vuka+ users and medical expert.
  Arms: Vuka+ App

SUMMARY:
This is a Type I Hybrid effectiveness-implementation trial to evaluate an HIV Pre-Exposure Prophylaxis (PrEP) medication adherence, persistence and social support app (Vuka+) for adolescent girls and young women (AGYW) in South Africa. This 6-month, 2-arm effectiveness and implementation trial (standard of care [SOC] vs. intervention app) will assess acceptability, feasibility and effectiveness. In addition, we will gather information on intervention delivery and barriers and facilitators for real-world delivery to inform future implementation and scale up.

DETAILED DESCRIPTION:
We will recruit 330 AGYW, aged 15-24 from the surrounding community, PrEP clinics and service providers in Cape Town, South Africa. If AGYW qualify for enrollment, they will be offered daily Truvada as PrEP. Participants will then be randomized 1:1 at baseline to SOC counselling and the Vuka+ intervention app or SOC counselling only (control). All participants will receive their regularly scheduled PrEP clinical care visits. At baseline, 1-, 3- and 6-month follow-up visits, participants will complete biobehavioral surveys, undergo HIV testing and pregnancy testing, and provide a urine (month 1 and 6) and DBS sample (months 1, 3 and 6) for tenofovir assessment. Intervention arm participants will also have the following study activities: install the intervention app on their phones at baseline study visit and be asked to use the intervention app for at least 5-10 minutes daily for 6 months. During this time, they will be prompted by the app to complete daily activities or health and wellness readings and to complete a weekly brief assessment related to their PrEP use. At follow-up study visits, intervention arm participants will complete an additional set of questions evaluating their app use experience and a subsample of participants will complete an in-depth qualitative exit interview to assess their app use experience, acceptability of the intervention and their evaluation of the app's content.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female at birth
* Age 15-24 years
* Healthy and weight at least 35kg
* Sexually active (had a male sexual partner in the past 6 months)
* Consistent access to a smartphone
* HIV-negative (clinic test)
* PrEP naive or no PrEP use in the past 6 months
* Eligible to start oral PrEP

Exclusion Criteria:

* Unable to currently start PrEP
* Abnormal laboratory, medical, physical, or social finding which could impact study participation, by investigator discretion
* Unwilling or unable to provide informed consent
* Participating in another PrEP trial
* Unwilling to provide at least 2 forms of contact for follow-up
* Taking renal toxic medications
* Sexual partner known to be HIV-positive

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 330 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
PrEP adherence | 3 months
  Adherence to PrEP was measured by tenofovir diphosphate (TFV-DP) concentrations in dried blood spots (DBS)

SECONDARY OUTCOMES:
Vuka+ app acceptability | 6 months
  Questionnaires and in-depth interviews were used to assess the acceptability of the smartphone app in the study population.
Vuka+ app usability | 6 months
  Quantitative self-reported usability measures (validated scales) were asked at follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Homaira Hanif, PhD, Principal Investigator — CONRAD/EVMS; Kathryn Muessig, PhD, Principal Investigator — FSU
Locations (1):
- Desmond Tutu Health Foundation, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No